CLINICAL TRIAL: NCT00184782
Title: Exploratory Study on FDG-PET Scanning in Evaluating the Metabolic Activity of Liver Metastases Before and After Resection of the Primary Tumor in Patients With a Colorectal Malignancy
Brief Title: Evaluation of Metabolic Activity of Liver Metastases by FDG-PET Scanning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CP 2005
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; liver metastases; metabolic activity
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Procedure: FDG-PET

SUMMARY:
The purpose of this study is to evaluate the effect of primary tumor resection on the metabolic activity of metastases in patients with a colorectal primary tumor and synchronous liver metastases by positron emission tomography (PET) with 2-deoxy-2-fluoro[18F]-D-glucose (FDG-PET) scanning.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the activity of liver metastases before and after resection of the primary tumor. Non-invasive assessment of tumor metabolism is possible in vivo by means of positron emission tomography (PET)-scanning. Therefore, FDG-PET scan offers a suitable approach to determine the influence of removal of a primary colorectal tumor on metabolic activity of the liver metastases. The FDG uptake in the liver metastases is quantified by calculating standardised uptake values (SUVs).

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer and synchronous liver metastases

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Increase in metabolic activity of liver metastases after resection of the primary tumor compared to the activity of metastases in patients without primary tumor resection

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands